CLINICAL TRIAL: NCT06714968
Title: The Effect of Digital Game on Assessing Nursing Students' Blood Pressure Measurement Skills
Acronym: DigitalGame
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanife DURGUN (Other)
Responsible Party: Sponsor-Investigator, Hanife DURGUN, Dr, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TABBO; Ordu University (Other Grant/Funding Number: Ordu University); B-2417 (Other Grant/Funding Number: Ordu University)
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Nursing Students
Keywords: Digital game, Nursing education,Blood pressure

STUDY DESIGN:
Intervention Model Description: This study was a randomized, single-blind, parallel group-controlled trial.
Who Masked: Participant
Masking Description: The study was single-blind and the participants were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control 1 (No Intervention): No intervention was applied to the students in the control group, and 2 weeks after the pre-test application, the post-test interface was activated for the students in this group and the students were enabled to perform the post-test application.
- control 2 (No Intervention): No intervention was applied to the students in the control group, and 2 weeks after the pre-test application, the post-test interface was activated for the students in this group and the students were enabled to perform the post-test application.
- Digital game (Experimental): After the pre-test application is completed, the students in the experimental group will be allowed to install the designed game application on their phones. After the installation process, students will be allowed to play the game for 2 weeks. After 2 weeks from the date of downloading the game, access to the game will be automatically blocked. After completing the application steps, when the student thinks that he/she is ready to apply the post-test, he/she will be able to perform the post-test application. In the post-test application, there will be no repeated return of the student to the questions or multiple answer submission. Two weeks after the application is completed, the knowledge test will be applied to the students again in order to objectively evaluate the learning. In this process, students will be prevented from accessing the application.
  Interventions: Other: Digital

INTERVENTIONS:
Other: Digital — After the pre-test application is completed, the students in the experimental group will be allowed to install the designed game application on their phones. After the installation process, students will be allowed to play the game for 2 weeks. After 2 weeks from the date of downloading the game, access to the game will be automatically blocked. After completing the application steps, when the student thinks that he/she is ready to apply the post-test, he/she will be able to perform the post-test application. In the post-test application, there will be no repeated return of the student to the questions or multiple answer submission. Two weeks after the application is completed, the knowledge test will be applied to the students again in order to objectively evaluate the learning. In this process, students will be prevented from accessing the application.
  Arms: Digital game

SUMMARY:
In recent years, in order for students to develop their skills related to the nursing profession, to cope with new and unpredictable clinical situations and to increase efficiency in nursing education, application contents such as simulation, video and mobile applications, in which students are active one-to-one and should take responsibility, rather than laboratory applications in which instructors are active, are developed to provide students with the opportunity to perform clinical nursing practices. Mobile applications, which are becoming increasingly popular in health education programmes and are also called e-health applications, are widely used and it is stated that they positively affect students' motivation and increase academic success. Although the use of games in nursing education dates back to the 1980s, the use of digital games in education is not very old, but it is an increasingly used teaching method in nursing practices that continue to develop. In addition, it is very important to use innovative learning strategies for new nurse candidates who are called Generation Z and who will soon become nursing professionals. Because, Generation Z is a generation born into the technology environment and actively uses this technology.

For this reason, in order to train nurses who are suitable and predisposed to the advancing technology, the nursing curriculum will ensure the support of the classroom and clinical environment, which will positively affect the quality and safety of patient care, and the organisation of a forward-looking, innovative and technology-oriented teaching curriculum will ensure the development of an easy and useful teaching method in teaching nursing practices.

Method: This study will be conducted in the form of an experimental design for first year nursing students in the period of February-March 2023.

DETAILED DESCRIPTION:
When the literature is examined, this study is a study that we want to pioneer a system that will contribute to the creation of an education curriculum that will help students who are generation Z and who will be the next professional nurses to learn more easily and effectively by using methods such as digital games before going to the clinical field by integrating the advancing technology and nursing practices into technology. Although the use of technology is currently used less or not at all in the education of individuals carrying out the nursing profession in clinics, the easier adaptation and use of new generation students to technology facilitates its use in nursing education. Therefore, the study was planned in the form of a digital game that students can adopt and apply more easily and quickly and at the same time to prevent errors in blood pressure application. As a result of this study, in addition to the teaching techniques in the nursing curriculum, a new curriculum that is more innovative and suitable for advancing technology will be adopted and will make a significant contribution to the implementation of nursing practices.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the research,
* Smartphone user,
* First year nursing student.
* Taking the Nursing Principles Course for the first time.

Exclusion Criteria:

* Graduated from health vocational high school,
* Previous knowledge of blood pressure measurement skills,
* Vertical transfer student,
* Wishing to leave the study at any stage of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Arterial Blood Pressure Academic Achievement Test | Immediately after randomisation (first measurement) 15 days later (2nd measurement) 1 month after randomisation (3rd measurement)
  The test prepared by Ziyai and Dikmen (2022) to test the level of knowledge about measuring arterial blood pressure consists of a total of 20 questions with five options. The questions in the test were prepared according to the level of the students and the suitability of the curriculum. The success score of the students was evaluated out of 100. In the study conducted by Ziyai and Dikmen, the internal consistency coefficient of the test was found to be 0.75.

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Durgun, Principal Investigator — Ordu University
Locations (1):
- Hanife Durgun, Ordu, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No